CLINICAL TRIAL: NCT06224192
Title: A Phase 3, Multicenter, Randomized, Open-label, Performance Study With Self-administered Subcutaneous Rocatinlimab (AMG 451) in Adolescent and Adult Subjects With Moderate-to-severe Atopic Dermatitis (AD) (ROCKET-Outpost)
Brief Title: A Study With Self-administered Rocatinlimab in Adolescent and Adult Participants With Moderate-to-severe Atopic Dermatitis
Acronym: ROCKET-Outpost
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230180
Record Dates: First submitted 2024-01-17; First posted 2024-01-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rocatinlimab Dose 1 Prefilled Syringe (PFS) (Experimental): Rocatinlimab will be self-administered subcutaneously using a PFS. Participants will receive rocatinlimab for 52 weeks.
  Interventions: Combination Product: Rocatinlimab Prefilled Syringe
- Rocatinlimab Dose 2 PFS (Experimental): Rocatinlimab will be self-administered subcutaneously using a PFS. Participants will receive rocatinlimab for 52 weeks.
  Interventions: Combination Product: Rocatinlimab Prefilled Syringe
- Rocatinlimab Dose 2 Autoinjector (AI) (Experimental): Rocatinlimab will be self-administered subcutaneously using an AI. Participants will received rocatinlimab for 52 weeks.
  Interventions: Combination Product: Rocatinlimab AI

INTERVENTIONS:
Combination Product: Rocatinlimab Prefilled Syringe — Prefilled Syringe (PFS) for subcutaneous (SC) injection self-administration of rocatinlimab.
  Other Names: AMG 451
  Arms: Rocatinlimab Dose 1 Prefilled Syringe (PFS); Rocatinlimab Dose 2 PFS
Combination Product: Rocatinlimab AI — AI for SC injection self-administration of rocatinlimab.
  Other Names: AMG 451
  Arms: Rocatinlimab Dose 2 Autoinjector (AI)

SUMMARY:
The primary objective of this study is to assess successful self-administration of rocatinlimab subcutaneously using devices for injection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 at Day 1.
* Diagnosis of AD according to American Academy of Dermatology (AAD) Consensus Criteria (2014) that has been present for at least 12 months.
* History of inadequate response to Topical Corticosteroids (TCS) of medium to higher potency (with or without topical calcineurin inhibitors [TCI]).
* Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD™) score ≥ 3 at screening and pre-randomization.
* Eczema Area and Severity Index (EASI) score ≥ 16 at initial at screening and pre-randomization.
* ≥ 10% body surface area (BSA) of AD involvement at screening and pre-randomization.

Exclusion Criteria:

* Treatment with a biological product within 12 weeks or 5 half-lives, whichever is longer, prior to day 1 pre-randomization.
* Treatment with any of the following medications or therapies within 5 half-lives prior to day 1 pre-randomization:

  1. Systemic corticosteroids
  2. Non-biologic, non-targeted systemic immunosuppressants
  3. Oral or Topical Janus kinase inhibitors
* Treatment with any of the following medications or therapies within 1 week before day 1 pre-randomization:

  1. Topical phosphodiesterase 4 (PDE4) inhibitors
  2. Other topical immunosuppressive agents (not including TCS/TCI)
  3. Combination topical agents containing any of the above components

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Proportion of Full-dose Self-administered Rocatinlimab Injections Among Total Attempted Injections up to Week 16 | Up to Week 16

SECONDARY OUTCOMES:
Proportion of Devices that Have Been Reported with Product Complaints Related to Function by Participants, Caregivers, or Investigators Among Total Dispensed Devices up to Week 16 | Up to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (47):
- United States (22):
  - Kern Research Inc, Bakersfield, California
  - Long Beach Research Institute, Long Beach, California
  - Dermatology Research Associates, Los Angeles, California
  - Havana Research Institute Inc, Pasadena, California
  - Integrative Skin Science and Research, Sacramento, California
  - Direct Helpers Research Center, Hialeah, Florida
  - Anchor Medical Research, Miami, Florida
  - Hamilton Research, LLC, Alpharetta, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Dermatology and Skin Cancer Center Leawood, Leawood, Kansas
  - Excel Clinical Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - The Skin Surgery Center for Clinical Research, Winston-Salem, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Apex Clinical Research Center LLC, Mayfield Heights, Ohio
  - Essential Medical Research LLC, Tulsa, Oklahoma
  - Health Concepts, Rapid City, South Dakota
  - Cumberland Skin Center, Hermitage, Tennessee
  - Sms Clinical Research Limited Liability Company, Mesquite, Texas
  - Texas Dermatology Research Center, Plano, Texas
  - Virginia Dermatology and Skin Cancer Center, Norfolk, Virginia
- Canada (11):
  - Interior Dermatology Centre, Kelowna, British Columbia
  - LEADER Research, Hamilton, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - DermEdge Research Incorporated, Mississauga, Ontario
  - Allergy Research Canada Incorporated, Niagara Falls, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - FACET Dermatology, Toronto, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - XLR8 Medical Research, Incorporated, Windsor, Ontario
  - Skinsense Medical Research, Saskatoon, Saskatchewan
- Japan (7):
  - Ekihigashi Dermatology Allergy Clinic, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Matsuo Clinic, Fukuoka, Fukuoka
  - Suizenji Dermatology Clinic, Kumamoto, Kumamoto
  - Dermatology and Ophthalmology Kume Clinic, Sakai-shi, Osaka
  - Mita Dermatology Clinic, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
- South Korea (7):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Ajou University Hospital, Suwon-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Guttman-Yassky E, Simpson E, Bissonnette R, Eichenfield LF, Kabashima K, Luna PC, Hercogova JT, Spelman L, Worm M, Esfandiari E, Arai T, Mano H, Charuworn P, Wang A, Kricorian G. ROCKET: a phase 3 program evaluating the efficacy and safety of rocatinlimab in moderate-to-severe atopic dermatitis. Immunotherapy. 2025 Feb;17(2):83-94. doi: 10.1080/1750743X.2025.2464528. Epub 2025 Feb 26. PMID 40012373
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com